CLINICAL TRIAL: NCT04646395
Title: Phase II Trial of Acalabrutinib in Combination With Tafasitamab in Patients With Previously Treated Marginal Zone Lymphomas (MZL)
Brief Title: Study of Acalabrutinib and Tafasitamab in MZL Patients
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: International Extranodal Lymphoma Study Group (IELSG) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IELSG49; 2019-004396-38 (EudraCT Number)
Record Dates: First submitted 2020-11-17; First posted 2020-11-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Marginal Zone Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone | interventions — tafasitamab; acalabrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tafasitamab and Acalabrutinib (Experimental): Acalabrutinib will be administered continuously at the dose of 100 mg BID (equivalent to a total daily dose of 200 mg), from day 1 to day 28 of each cycle for 24 cycles.
  Tafasitamab will be administered 12 mg/kg iv on days 1, 8, 15 and 22 for the first 3 cycles. Then patients will continue treatment until cycle 24 with tafasitamab 12mg/kg iv on day 1
  Interventions: Drug: Tafasitamab; Drug: Acalabrutinib

INTERVENTIONS:
Drug: Tafasitamab — 200 mg powder for reconstitution with 5 ml water for injection
  Other Names: MOR00208
Drug: Acalabrutinib — 100 mg hard gelatin capsules
  Other Names: Calquence

SUMMARY:
This is a multicenter open label phase II trial in patients with previously treated Marginal Zone Lymphomas.

The aim of the study is to evaluate the efficacy and the safety of tafasitamab in combination with acalabrutinib.

Twenty-four patients are expected to be enrolled and treated every 28 days with acalabrutinib and tafasitamab for 24 cycles.

The study consists of two parts, which are performed sequentially. The first part is a safety run-in to evaluate the safety data once 6 patients (representing the 25% of the total cohort) have completed the first cycle of treatment. An Independent Data Monitoring Committee (IDMC) will provide an independent assessment of this evaluation.

The second part starts after the outcome of this evaluation and will include the remaining 18 patients. The 6 patients of the safety run-in phase will be considered for the final evaluation of the study.

Between 11 - 13 weeks, patients showing partial or complete response (PR, CR) will continue treatment, while patients showing stable disease (SD) will discontinue it. However, patients in SD who benefit from therapy may continue to be treated, after agreement between the Investigator and the Sponsor.

Patients who complete the 24 cycles of treatment will enter the follow-up phase up to 3 years from patient's last study treatment dose (about 5 years from treatment start).

Patients who discontinue treatment before cycle 24 for any reason will be followed for up to 3 years (every 6 months for the first year and yearly for the second and third year) from the patient's last study treatment dose.

.

DETAILED DESCRIPTION:
Marginal zone B cell lymphomas (MZLs) comprise three distinct entities: extranodal MZL (EMZL) of mucosa-associated lymphoid tissue type (MALT) lymphoma, splenic MZL (SMZL) and nodal MZL (NMZL).

Together they represent approximately 5%-15% of all non-Hodgkin lymphomas.

MZL are in general indolent lymphomas with relatively low risk of transformation. The available treatment options can lead to responses but disease recurrence is often observed. For patients with MZL and recurrent disease following initial treatment, currently there is no established standard therapy and new treatment options and treatment combinations are needed.

The proposed trial will evaluate the safety and efficacy of the anti-CD19 monoclonal antibody tafasitamab in combination with the BTK inhibitor acalabrutinib. The B-lymphocyte, lineage specific surface antigen CD19 is broadly and homogeneously expressed in MZLs. This makes CD19 an attractive target for the treatment of MZL patients, in particular those who failed a previous rituximab-containing regimen.

On the other hand, genetic and immunogenetic data point to B-cell receptor signalling as a key oncogenic pathway of MZLs. The activity of single agent ibrutinib in MZLs is an in vivo proof that MZLs are addicted of BTK-driven signalling and that the BCR pathway is a vulnerability of these lymphomas.

The safety profile of the anti CD19 monoclonal antibody tafasitamab and of the BTK inhibitor acalabrutinib indicate the possibility that their combination can be developed without major overlapping side effects.

The proposed trial is a prospective multicenter trial combining tafasitamab and acalabrutinib in patients with MZL (including EMZL, SMZL and NMZL) with disease refractory to or in first or greater relapse after prior systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and willingness to sign a written informed consent
* Histologically confirmed diagnosis of MZL.
* Disease refractory to or in first or greater relapse after prior systemic therapy.
* In need of treatment disease satisfying the following criteria:

  * EMZL: symptomatic lymphoma or with other treatment indications (overt progression, deep invasion, bulky disease, impending organ damage, patient preference), symptomatic disseminated disease, contraindications to RT, failure after antibiotics or after local therapy,
  * SMZL: presence of progressive or symptomatic splenomegaly and/ or any progressive cytopaenias,
  * NMZL: B symptoms, deterioration of peripheral blood counts due to lymphoma infiltration of the bone marrow, rapid enlargement of lymph nodes or compression of vital organs by bulky disease.
* Measurable or non-measurable lesions where the response is nevertheless evaluable by non-imaging means (e.g., gastric or bone marrow infiltrations).
* Ann Arbor Stage I-IV.
* ECOG performance status of 0, 1 or 2 with no deterioration over the previous 2 weeks prior to registration .
* Age ≥ 18 years.
* Absolute neutrophil count (ANC) ≥ 1.000/mm3 and platelets ≥ 100.000/mm3, unless these abnormalities are related to bone marrow infiltration or to hypersplenism.
* Adequate hepatic function, renal function and coagulation parameters
* Women with childbearing potential who are using highly effective contraception, are not pregnant or lactating and agree not to become pregnant during trial treatment and for at least 3 months after the last IMP dose.
* Men who agree not to father a child during trial treatment and for at least 3 months after the last IMP dose.
* Patient able and willing to swallow trial drugs as whole capsule

Exclusion Criteria:

* History of prior malignancy that could affect compliance with the protocol or interpretation of results, except for the following:

  1. Curatively treated basal cell carcinoma or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or carcinoma in situ of the prostate at any time prior to study,
  2. Other cancers not specified above that have been curatively treated by surgery and/or radiation therapy from which patient is disease-free for ≥3 years without further treatment.
* Major surgery and any systemic anti-cancer treatment within 3 weeks prior to registration.
* Prior exposure to a BTK inhibitor or CD19-targeted therapy.
* Steroid therapy for anti-neoplastic intent.
* Severe or uncontrolled cardiovascular disease
* History of cerebrovascular accident or intracranial hemorrhage within 6 months prior to registration and known bleeding disorders
* Patients with a history of confirmed progressive multifocal leukoencephalopathy (PML).
* Concomitant diseases that require anticoagulant therapy with warfarin or phenoprocoumon or other vitamin K antagonists and patients treated with dual anti-platelet therapy. Patients being treated with factor Xa inhibitors (e.g. rivaroxaban, apixaban, edoxaban), direct thrombin inhibitors (e.g. dabigatran) LMWH, or single anti-platelets agents (e.g. aspirin, clopidogrel) can be included, but must be properly informed about the potential risk of bleeding.
* Malabsorption syndrome or other condition that precludes enteral route of administration.
* Active human immunodeficiency virus (HIV) or active chronic hepatitis C or hepatitis B virus infection or any uncontrolled active systemic infection requiring intravenous (iv) antimicrobial treatment.
* Active, uncontrolled autoimmune phenomenon (autoimmune hemolytic anemia or immune. thrombocytopenia) requiring steroid therapy with > 20 mg daily of prednisone dose or equivalent.
* Known hypersensitivity to trial drugs or to any component of the trial drugs.
* Concomitant treatment with strong CYP3A inducers or inhibitors
* Treatment with proton pump inhibitors. Subjects receiving proton pump inhibitors who switch to antacids are eligible for enrollment to this study.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that in the opinion of the investigator may increase the risk associated with trial participation or IMPs administration or may interfere with the interpretation of trial results and/or would make the patient inappropriate for enrolment into this trial.
* Concurrent participation in another therapeutic clinical trial
* History of or ongoing confirmed central nervous system (CNS) lymphoma
* Patients who received any IMP within 30 days or 5 half-lives (whichever is shorter) before the first dose of the study IMP
* Pregnant or breastfeeding women
* Patients who received a live virus vaccination within 28 days of the first IMP dose

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2027-09-15 (Estimated); Study Completion 2028-03-15 (Estimated)

PRIMARY OUTCOMES:
Complete Response (CR) Rate as best response to treatment | Between 11 - 13 weeks after treatment start, at the end of cycles 6, 12, 18, 24 (each cycle is 28 days)
  defined according to the international Revised Response Criteria for Malignant Lymphoma (Cheson et al 2014). For patients with SMZL, response is defined according to Matutes et al. 2008 and for patients with gastric lymphomas, histological response is evaluated according to GELA scoring system (Copie-Bergman et al 2003).

SECONDARY OUTCOMES:
Number of treatment emergent adverse events (AE) | From the time of informed consent signature until 28 days after treatment discontinuation or until resolution of all treatment-related AEs, whichever occurs later.
  Analysis of type and severity of Adverse Events according to CTCAE v5.0 and relationship to study treatment
Overall Response Rate (ORR) | Between 11 - 13 weeks after treatment start, at the end of cycles 6, 12, 18, 24 (each cycle is 28 days)
  ORR will be defined as sum of PR plus CR defined according to the revised response criteria for malignant lymphomas (Cheson et al 2014), to the GELA Histological Grading System for gastric EMZL and the Matutes criteria for SMZL.
Progression Free Survival (PFS) | From the date of treatment start to the date of progression or the date of death for any cause until 3 years from last treatment dose
  PFS will be computed from the first IMP dose to date of disease progression or date of death for any reason or censored at the date of the last follow-up visit, whichever occurs earlier
Duration of response (DoR) | From the date of the first documented response to the date of disease progression or relapse or death until 3 years from last treatment dose
  DOR will be define as the time between the first documented response to therapy and subsequent disease progression or relapse or death according to the international Revised Response Criteria for Malignant Lymphoma (Cheson et al 2014).
Overall Survival (OS) | From the date of treatment start to the date of death for any cause until 3 years from last treatment dose
  Overall survival (OS) will be computed from the first IMP dose to the date of death for any reason or censored at the date of the last contact, whichever occurs earlier

CONTACTS AND LOCATIONS:
Overall Officials: Anastasios Stathis, MD, Study Chair — Oncology Institute of Southern Switzerland - Bellinzona, Switzerland; Davide Rossi, MD, Study Chair — Oncology Institute of Southern Switzerland - Bellinzona, CH; Emanuele Zucca, MD, Study Chair — Oncology Institute of Southern Switzerland - Bellinzona, CH
Locations (9):
- University of Wien, Vienna, Austria
- Italy (7):
  - ASST Spedali Civili di Brescia, Brescia
  - Fondazione IRCCS - Istituto Nazionale dei Tumori, Milan
  - Fondazione IRCCS Cà Granda-Ospedale Maggiore Policlinico, Milan
  - Ospedale Maggiore della Carità, Novara
  - AUSL Ravenna U.O. Ematologia, Ravenna
  - Azienda Ospedaliera - IRCCS - Arcispedale Santa Maria Nuova, Reggio Emilia
  - Ospedale di Circolo e Fondazione Macchi - ASST Sette Laghi, Varese
- Oncology Institute of Southern Switzerland, Bellinzona, Switzerland